CLINICAL TRIAL: NCT01722292
Title: A Phase 1b/2 Double-Blind Randomized Trial of the Hedgehog/SMO Antagonist LY2940680 in Combination With Carboplatin and Etoposide Followed by LY2940680 Versus Carboplatin and Etoposide Plus Placebo Followed by Placebo in Patients With Extensive-Stage Small Cell Lung Cancer
Brief Title: A Study of LY2940680 in Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Change in clinical strategy.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14631; I4J-MC-HHBE (Other: Eli Lilly and Company); 2012-003174-83 (EudraCT Number)
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2015-09

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — LY2940680; Carboplatin; Etoposide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1b: LY2940680 + C + E (Experimental): Phase 1b Dose Escalation: Cycles 1-6 (21 day cycles) LY2940680 administered orally, once daily at escalating doses (100 milligrams [mg] up to 400 mg) in combination with etoposide (E) 100 milligram per square meter (mg/m^2) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle and carboplatin (C) Area Under the Curve [AUC] 5 (mg•min/mL) administered by IV infusion on day 1 each cycle.
  Phase 1b Maintenance: Cycles 7+ (21 day cycles) LY2940680 administered orally, once daily at the same dose as induction. Participants receiving benefit may continue until disease progression, unacceptable toxicity, or discontinuation.
  Interventions: Drug: LY2940680; Drug: Carboplatin; Drug: Etoposide
- Phase 2: Placebo + C + E (Placebo Comparator): Induction: Cycles 1-6 (21 day cycles) Placebo administered orally once daily in combination with etoposide 100 mg/m2 administered by IV infusion on days 1, 2, 3 of each cycle and carboplatin AUC 5 administered by IV infusion on day 1 each cycle.
  Maintenance: Cycles 7+ (21 day cycles) Placebo administered orally once daily. Participants receiving benefit may continue until disease progression, unacceptable toxicity, or discontinuation.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Placebo
- Phase 2: LY2940680 + C+ E (Experimental): Induction: Cycles 1-6 (21 day cycles) LY2940680 (dose to be determined in Phase 1b portion) administered orally once daily in combination with etoposide 100 mg/m^2 administered by IV infusion on days 1, 2, 3 of each cycle and carboplatin AUC 5 administered by IV infusion on day 1 each cycle.
  Maintenance: Cycles 7+ (21 day cycles). LY2940680 (dose to be determined in Phase 1 portion) administered orally once daily.
  Interventions: Drug: LY2940680; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: LY2940680 — Administered orally
  Arms: Phase 1b: LY2940680 + C + E; Phase 2: LY2940680 + C+ E
Drug: Carboplatin — Administered IV
Drug: Etoposide — Administered IV
Drug: Placebo — Administered orally
  Arms: Phase 2: Placebo + C + E

SUMMARY:
The purpose of this study is to find a recommended dose of LY2940680 that can be safely given in combination with etoposide and carboplatin followed by LY2940680 alone in participants with extensive-disease small cell lung cancer. The study will also compare progression-free survival in participants who are administered etoposide, carboplatin and LY2940680 followed by LY2940680 alone versus etoposide, carboplatin, and placebo followed by placebo alone.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of Small Cell Lung Cancer (SCLC), including malignant pleural effusion that is extensive stage per the International Staging System
* Performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) performance status schedule
* No prior systemic chemotherapy, immunotherapy, or biological therapy for SCLC
* Prior radiation therapy allowed to <25% of the bone marrow. Participants who have received prior radiation to the whole pelvis or chest for the treatment of SCLC are not eligible
* At least 1 unidimensionally measurable lesion meeting Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Adequate organ function including the following:

  * Adequate bone marrow reserve: absolute neutrophil count (ANC) ≥1.5 x 10^9/ liter (L), platelets ≥100 x 10^9/L, and hemoglobin ≥9 grams/deciliter (g/dL)
  * Hepatic: bilirubin ≤1.5 times the upper limit of normal (ULN), alkaline phosphatase (AP), Serum alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤3.0 x ULN (AP, AST, and ALT ≤5 x ULN is acceptable if liver has tumor involvement)
  * Renal: calculated creatinine clearance (CrCl) ≥50 milliliters per minute (mL/min) based on the standard Cockcroft and Gault formula
* Estimated life expectancy of at least 12 weeks
* For women: Must be surgically sterile, post-menopausal, or compliant with a medically approved contraceptive regimen during and for 6 months after the treatment period; must have a negative serum pregnancy test within 7 days before study enrollment. For men: Must be surgically sterile or compliant with a contraceptive regimen during and for 6 months after the treatment period
* Availability of a tumor tissue sample
* Able to swallow capsules

Exclusion Criteria:

* Currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have previously participated in a study involving LY2940680
* Have previously received treatment with carboplatin or etoposide
* Have a mixed histological diagnosis of SCLC and Non-Small Cell Lung Cancer (NSCLC)
* Have a serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the participant's ability to adhere to the protocol
* Have an active infection [≥38.5 degrees Celsius and/or receiving Intravenous (IV) antibiotic therapy]
* Have a serious cardiac condition
* Have had a prior malignancy other than SCLC, carcinoma in situ of the cervix, or nonmelanoma skin cancer, unless that prior malignancy was diagnosed and definitively treated at least 5 years previously with no subsequent evidence of recurrence. Participants with a history of non-metastatic prostate cancer, including biochemical relapse only, will be eligible even if diagnosed less than 5 years previously
* Symptomatic central nervous system (CNS) metastases and asymptomatic CNS metastases requiring concurrent corticosteroid therapy. Treated stable CNS metastases are allowed; the participant must be stable after radiotherapy for ≥2 weeks and off of corticosteroids for ≥1 week
* Presence of clinically significant third-space fluid collections that cannot be controlled prior to study entry
* Significant weight loss (that is, ≥10%) over the 6-week period prior to study entry
* Concurrent administration of any other antitumor therapy. An exception will be made for non-metastatic prostate cancer participants continuing androgen blockade therapy only or breast cancer participants continuing adjuvant antiestrogen therapy only (for example, an aromatase inhibitor)
* Females who are breastfeeding
* Have corrected QT interval (QTc) of >470 millisecond (msec) on screening electrocardiogram (ECG)
* Have received medications that are strong inhibitors of Cytochrome P450 3A4 (CYP3A4) within 7 days prior to receiving study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (12):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology Associate, Albany, New York
  - Mount Sinai Medical Center, New York, New York
  - Clinical Research Unit (ITOR) Greenville Hospital System, Greenville, South Carolina
  - Accelerated Comm. Oncology Research Network (ACORN), Memphis, Tennessee
  - The West Clinic, Memphis, Tennessee
  - US Oncology, The Woodlands, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Northwest Cancer Specialists PC, Vancouver, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
- United Kingdom (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to strategic reasons, the Phase 2 portion was not initiated, and further clinical development was stopped. Phase 1b study completer was defined as completion of the dose-limiting toxicity (DLT) period (1 cycle- 21 days cycle for LY2940680 in combination with carboplatin and etoposide.
Groups:
- Phase 1b: 100 mg LY2940680 + C + E: 100 milligrams (mg) LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve (AUC) 5 milligrams*minute*milliliters (mg•min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
  Maintenance:
  Single-agent LY2940680 administered orally QD at the same dose as induction at Cycles 7+ (21 day cycles). Participants receiving benefit may continue until disease progression, unacceptable toxicity, or discontinuation.
- Phase 1b: 200 mg LY2940680 + C + E: 200 mg LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve (AUC) 5 milligrams*minute*milliliters (mg•min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
  Maintenance:
  Single-agent LY2940680 administered orally QD at the same dose as induction at Cycles 7+ (21 day cycles). Participants receiving benefit may continue until disease progression, unacceptable toxicity, or discontinuation.
- Phase 1B: 400 mg LY2940680 + C + E: 400 mg LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve (AUC) 5 milligrams*minute*milliliters (mg•min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
  Maintenance:
  Single-agent LY2940680 administered orally QD at the same dose as induction at Cycles 7+ (21 day cycles). Participants receiving benefit may continue until disease progression, unacceptable toxicity, or discontinuation.
Period: Overall Study
Arm/Group | Phase 1b: 100 mg LY2940680 + C + E | Phase 1b: 200 mg LY2940680 + C + E | Phase 1B: 400 mg LY2940680 + C + E
Started | 6 | 6 | 14
Received at Least One Dose of Study Drug | 6 | 6 | 14
Completed | 6 | 6 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Phase 1b: 100 mg LY2940680 + C +E: 100 mg LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 milligrams*minute*milliliters (mg•min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
  Maintenance:
  Single-agent LY2940680 administered orally QD at the same dose as induction at Cycles 7+ (21 day cycles). Participants receiving benefit may continue until disease progression, unacceptable toxicity, or discontinuation.
- Phase 1b: 200 mg LY2940680 + C + E: 200 mg LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 milligrams*minute*milliliters (mg•min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
  Maintenance:
  Single-agent LY2940680 administered orally QD at the same dose as induction at Cycles 7+ (21 day cycles). Participants receiving benefit may continue until disease progression, unacceptable toxicity, or discontinuation.
- Phase 1b: 400 mg LY2940680 + C + E: 400 mg LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 milligrams*minute*milliliters (mg•min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
  Maintenance:
  Single-agent LY2940680 administered orally QD at the same dose as induction at Cycles 7+ (21 day cycles). Participants receiving benefit may continue until disease progression, unacceptable toxicity, or discontinuation.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: 100 mg LY2940680 + C +E | Phase 1b: 200 mg LY2940680 + C + E | Phase 1b: 400 mg LY2940680 + C + E | Total
Number analyzed (Participants) | 6 | 6 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.35) | 64.8 (11.96) | 60.2 (12.19) | 62.2 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 7 | 13
  Male | 3 | 3 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 5 | 14 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 6 | 3 | 13 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10 | 20
  United Kingdom | 1 | 1 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Recommended Phase 2 Dose of LY2940680: Maximum Tolerated Dose (MTD)
Description: MTD was defined as the highest tested dose that has <33% probability of causing a dose-limiting toxicity(DLT). DLT was defined as an AE during Cycle 1 that is possibly related to the study drug and fulfills any one of the following criterion using the National Cancer Institute(NCI) Common Terminology Criteria for Adverse Events(CTCAE),version 4.0:Grade 3 non-hematological toxicity except nausea, vomiting, constipation, diarrhea, fatigue, or anorexia that is manageable with appropriate care,transient(i.e., ≤5 days) Grade 3 elevations of alanine aminotransferase(ALT) and/or aspartate aminotransferase(AST), without evidence of other hepatic injury, in the setting of preexisting hepatic metastasis, ≥Grade 3 thrombocytopenia with bleeding or Grade 4 thrombocytopenia of any duration,CTCAE Grade 4 hematological toxicity of >5 days duration and any febrile neutropenia. any other significant toxicity deemed by the primary investigator and Lilly clinical research personnel to be dose-limiting.
Time Frame: Baseline to Completion of the Phase 1b (Up To 12 Months)
Population: All participants who received at least one dose of study drug and were enrolled in Phase1b of the study.
Measure: Number; unit: milligrams (mg)
Groups:
- Phase 1b: Cohort 1:
  100 milligrams (mg) LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg*min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
  Cohort 2:
  200 milligrams (mg) LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg*min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
  Cohort 3:
  400 milligrams (mg) LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg*min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
Arm/Group | Phase 1b
Number analyzed (Participants) | 26
milligrams (mg) | 400

2. Primary Outcome: Phase 2: Progression-Free Survival
Time Frame: Randomization to Measured Progressive Disease or Death of Any Cause (Estimated as 18 Months)
Population: Zero participants analyzed. Due to strategic reasons, the Phase 2 portion was not initiated, and further clinical development was stopped.
Groups:
- Phase 2: 400 mg LY2940680 + C+ E: 400 mg LY2940680 administered orally QD cycles 1-6 (21 day cycle).
  (AUC) 5 carboplatin (C) administered by IV infusion on day 1 each cycle.
  100 mg/m^2 etoposide (E) administered by IV infusion on days 1, 2, 3 of each cycle, followed by a single agent of LY2940680.
- Phase 2: Placebo + C + E: Placebo administered orally QD for 6 cycles.
  (AUC) 5 carboplatin administered by IV infusion on day 1 of each cycle.
  100 mg/m^2 etoposide administered by IV infusion on days 1, 2, 3 of each cycle.
Arm/Group | Phase 2: 400 mg LY2940680 + C+ E | Phase 2: Placebo + C + E
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Phase 1b and 2: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY2940680, LSN3185556 at the Recommended Dose
Time Frame: Cycle (C)1 Day (D) 1:Predose,0.5 ,1, 2, 4, 6, 8h; C2 D1:Pr,0.5,1,2,4,6,8 hours
Population: All participants who received at least one dose of study drug and were enrolled in Phase 1b study. Due to strategic reasons, the Phase 2 portion was not initiated, and further clinical development was stopped.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Groups:
- Phase 1b: 100 mg LY2940680 + C + E: 100 mg LY2940680 administered orally once daily (QD) for 6 cycles.
  100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg*min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
- Phase 1b: 200 mg LY2940680 + C + E: 200 mg LY2940680 administered orally once daily (QD) for 6 cycles.
  100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg*min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
- Phase 1B: 400 mg LY2940680 + C + E: 400 mg LY2940680 administered orally once daily (QD) for 6 cycles.
  100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg*min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
Arm/Group | Phase 1b: 100 mg LY2940680 + C + E | Phase 1b: 200 mg LY2940680 + C + E | Phase 1B: 400 mg LY2940680 + C + E
Number analyzed (Participants) | 6 | 6 | 14
microgram per milliliter (µg/mL)
  LY2940680 Cycle 1, Day 1 | 0.491 (64) | 1.01 (36) | 1.56 (35)
  LY2940680 Cycle 2, Day 1 | 0.578 (71) | 1.16 (66) | 3.29 (33)
  LSN3185556 Cycle 1, Day 1 | 0.444 (33) | 0.737 (138) | 1.75 (47)
  LSN3185556 Cycle 2, Day 1 | 1.6 (35) | 2.1 (90) | 6 (59)

4. Secondary Outcome: Phase 1b and 2: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Carboplatin and Etoposide at the Recommended Dose
Time Frame: Cycle (C)1 Day (D) 1:Predose,0.5 ,1, 2, 4, 6, 8h; C2 D1:Pr,0.5,1,2,4,6,8 hours
Population: All participants who received at least one dose of study drug and were enrolled in Phase 1b study. Due to strategic reasons, the Phase 2 portion was not initiated, and further clinical development was stopped.
  C and E doses did not change for the 3 cohorts of LY (100,200 and 400 mg) so we only need to report one grouping.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Groups:
- Phase 1b: LY2940680 + C + E: LY2940680 administered orally once daily (QD) for 6 cycles.
  100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg*min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
Arm/Group | Phase 1b: LY2940680 + C + E
Number analyzed (Participants) | 26
microgram per milliliter (µg/mL)
  Total Carboplatin Cycle 1, Day 1 | 16.7 (33)
  Total Carboplatin Cycle 2, Day 1 | 13.1 (42)
  Etoposide Cycle 1, Day 1 | 20.9 (18)
  Etoposide Cycle 2, Day 1 | 18.4 (28)

5. Secondary Outcome: Phase 1b and 2: Pharmacokinetics: Area Under the Curve ( AUC₀-₂₄) for LY2940680 and LSN3185556 at the Recommended Dose
Time Frame: Cycle (C)1 Day (D) 1:Predose,0.5 ,1, 2, 4, 6, 8h; C2 D1:Pr,0.5,1,2,4,6,8 hours
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per milliliter (h.µg/mL)
Groups:
- Phase 1b: 100 mg LY2940680 + C+ E: 100 mg LY2940680 administered orally once daily (QD) for 6 cycles.
  100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg*min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
- Phase 1b: 200 mg LY2940680 + C+ E: 200 mg LY2940680 administered orally once daily (QD) for 6 cycles.
  100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg*min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
- Phase 1b: 400 mg LY2940680 + C+ E: 400 mg LY2940680 administered orally once daily (QD) for 6 cycles.
  100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg*min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
Arm/Group | Phase 1b: 100 mg LY2940680 + C+ E | Phase 1b: 200 mg LY2940680 + C+ E | Phase 1b: 400 mg LY2940680 + C+ E
Number analyzed (Participants) | 6 | 6 | 14
Hour*microgram per milliliter (h.µg/mL)
  LY2940680 Cycle 1, Day 1 | 6.34 (57) | 8.96 (39) | 15.9 (27)
  LY2940680 Cycle 2, Day 1 | 7.86 (67) | 15.5 (64) | 37.6 (43)
  LSN3185556 Cycle 1, Day 1 | 7.23 (49) | 16.2 (67) | 26 (37)
  LSN3185556 Cycle 2, Day 1 | 22.7 (58) | 31.1 (111) | 92.5 (72)

6. Secondary Outcome: Phase 1b and 2: Pharmacokinetics: Area Under the Curve ( AUC₀-₂₄) for Etoposide and as AUC₀-₆ for Carboplatin at the Recommended Dose
Time Frame: Cycle (C)1 Day (D) 1:Predose,0.5 ,1, 2, 4, 6, 8h; C2 D1:Pr,0.5,1,2,4,6,8 hours
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per milliliter (h.µg/mL)
Groups:
- Phase 1b: LY2940680 + C+ E: LY2940680 administered orally once daily (QD) for 6 cycles.
  100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg*min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
Arm/Group | Phase 1b: LY2940680 + C+ E
Number analyzed (Participants) | 26
Hour*microgram per milliliter (h.µg/mL)
  Total Carboplatin Cycle 1, Day 1 | 37.2 (23)
  Total Carboplatin Cycle 2, Day 1 | 32.0 (25)
  Etoposide Cycle 1, Day 1 | 104 (22)
  Etoposide Cycle 2, Day 1 | 96.1 (20)

7. Secondary Outcome: Phase 1b: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Overall Response Rate [ORR])
Description: ORR was defined as the percentage of all randomized participants with the best overall response of PR or CR using Response Evaluation Criteria in Solid Tumors (RECIST v1.1). CR is the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Tumor marker results must have normalized. PR is at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline to Study Completion Up to 39 Months
Population: All participants who received at least one dose of drug.
Measure: Mean (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b: 100 mg LY2940680 + C+ E | Phase 1b: 200 mg LY2940680 + C+ E | Phase 1b: 400 mg LY2940680 + C+ E
Number analyzed (Participants) | 6 | 6 | 14
percentage of participants | 50 [16.4 to 83.6] | 50 [16.4 to 83.6] | 57.1 [35.4 to 78.9]

8. Secondary Outcome: Phase 1b: Percentage Inhibition of Expression Levels of Gli1 in Skin Cells
Description: The gene expression data (Gli1) was normalized and the level of percentage of Gli1 inhibition post treatment was calculated.
Time Frame: Baseline, Cycle 2 Day 1, Cycle 7 Day 1
Population: All participants who received at least one dose of drug and had samples available.
Measure: Median (Inter-Quartile Range); unit: Percentage of Gli 1 Inhibition
Groups:
- Phase 1b: 100 mg LY2940680: 100 mg LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg*min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
- Phase 1b: 200 mg LY2940680: 200 mg LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg*min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
- Phase 1b: 400 mg LY2940680: 400 mg LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg*min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
Arm/Group | Phase 1b: 100 mg LY2940680 | Phase 1b: 200 mg LY2940680 | Phase 1b: 400 mg LY2940680
Number analyzed (Participants) | 5 | 5 | 12
Percentage of Gli 1 Inhibition | 94.7 [75.9 to 94.9] | 95.1 [94.5 to 97.2] | 94.8 [90.7 to 97.3]

9. Secondary Outcome: Phase 2: Overall Survival
Time Frame: Randomization to Study Completion (Estimated as 38 Months)
Population: as for outcome 2
Groups:
- Phase 2: 400 mg LY2940680 + C+ E: 400 mg LY2940680 administered orally QD cycles 1-6 (21 day cycle)
  (AUC) 5 carboplatin (C) administered by IV infusion on day 1 each cycle.
  100 mg/m^2 etoposide (E) administered by IV infusion on days 1, 2, 3 of each cycle, followed by a single agent of LY2940680.
Arm/Group | Phase 2: 400 mg LY2940680 + C+ E | Phase 2: Placebo + C + E
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Phase 2: Percent Change in Tumor Size (CTS)
Time Frame: Randomization to End of Cycle 2 (Estimated as 24 Months)
Population: as for outcome 2
Arm/Group | Phase 2: 400 mg LY2940680 + C+ E | Phase 2: Placebo + C + E
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Phase 2: Number of Participants With a Complete or Partial Tumor Response (Overall Response Rate)
Time Frame: Randomization to Study Completion (Estimated as 38 Months)
Population: as for outcome 2
Groups:
- Phase 2: Placebo + C + E: Induction: Cycles 1-6 (21 day cycles) Placebo administered orally once daily in combination with etoposide 100 mg/m^2 administered by IV infusion on days 1, 2, 3 of each cycle and carboplatin AUC 5 administered by IV infusion on day 1 each cycle.
  Maintenance: Cycles 7+ (21 day cycles) Placebo administered orally once daily. Participants receiving benefit may continue until disease progression, unacceptable toxicity, or discontinuation.
Arm/Group | Phase 2: Placebo + C + E | Phase 2: LY2940680 + C+ E
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Phase 1b and 2: Pharmacokinetics: Time to Maximal Concentration (Tmax) of LY2940680 andLSN3185556 at the Recommended Dose
Time Frame: Cycle (C)1 Day (D) 1:Predose,0.5 ,1, 2, 4, 6, 8h; C2 D1:Pr,0.5,1,2,4,6,8 hours
Population: as for outcome 3
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Phase 1b: 100 mg LY2940680 + C+ E | Phase 1b: 200 mg LY2940680 + C+ E | Phase 1b: 400 mg LY2940680 + C+ E
Number analyzed (Participants) | 6 | 6 | 14
Hour (h)
  LY2940680 Cycle 1, Day 1 | 2.05 [1 to 3.98] | 2.01 [1.03 to 2.05] | 1.51 [0.5 to 6]
  LY2940680 Cycle 2, Day 1 | 2.96 [0.08 to 5.83] | 4 [1.88 to 4.08] | 1 [0.5 to 6]
  LSN3185556 Cycle 1, Day 2 | 6.14 [2 to 24.03] | 5.87 [2.07 to 24.97] | 6 [2.05 to 24]
  LSN3185556 Cycle 2, Day 2 | 2.3 [0 to 4] | 4.08 [4 to 23.83] | 2.21 [0.5 to 6]

13. Secondary Outcome: Phase 1b and 2: Pharmacokinetics: Time to Maximal Concentration (Tmax) of Carboplatin and Etoposide at the Recommended Dose
Time Frame: Cycle (C)1 Day (D) 1:Predose,0.5 ,1, 2, 4, 6, 8h; C2 D1:Pr,0.5,1,2,4,6,8 hours
Population: as for outcome 4
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Phase 1b: LY2940680 + C+ E
Number analyzed (Participants) | 26
Hour (h)
  Total Carboplatin Cycle 1, Day 1 | 0.5 [0.42 to 1.08]
  Total Carboplatin Cycle 2, Day 1 | 0.5 [0.42 to 1.05]
  Etoposide Cycle 1, Day 1 | 0.96 [0.48 to 1.5]
  Etoposide Cycle 2 ,Day 1 | 0.99 [0.33 to 1.17]

ADVERSE EVENTS:
Groups:
- Phase 1b: 100 mg LY2940680 + C + E: 100 mg LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg•min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
- Phase 1b: 200 mg LY2940680 + C + E: 200 mg LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg•min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
- Phase 1b: 400 mg LY2940680 + C + E: 400 mg LY2940680 administered orally once daily (QD) for 6 cycles. 100 mg per square meter (mg/m^2) etoposide (E) administered by intravenous (IV) infusion on days 1, 2, 3 of each cycle.
  Area under the Curve [AUC] 5 (mg•min/mL) carboplatin (C) administered by IV infusion on day 1 each cycle.
Arm/Group | Phase 1b: 100 mg LY2940680 + C + E | Phase 1b: 200 mg LY2940680 + C + E | Phase 1b: 400 mg LY2940680 + C + E
Serious Adverse Events (participants affected / at risk) | 3/6 | 6/6 | 8/14
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: 100 mg LY2940680 + C + E (N=6) | Phase 1b: 200 mg LY2940680 + C + E (N=6) | Phase 1b: 400 mg LY2940680 + C + E (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase 1b: 100 mg LY2940680 + C + E (N=6) | Phase 1b: 200 mg LY2940680 + C + E (N=6) | Phase 1b: 400 mg LY2940680 + C + E (N=14)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 3 (5) | 8 (12)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (9) | 5 (8) | 7 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (6) | 3 (3) | 8 (14)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (11)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (5) | 10 (13)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (5) | 4 (6) | 5 (9)
Asthenia (General disorders) | 1 (1) | 2 (2) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 3 (3) | 11 (15)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 4 (4) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (2) | 1 (2)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 6 (7)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (3) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3) | 6 (7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 3 (4)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (4) | 4 (4) | 8 (9)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1/7 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 7 (7)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to strategic reasons, the Phase 2 portion was not initiated, and further clinical development was stopped.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days